CLINICAL TRIAL: NCT01258907
Title: A Multicenter, Randomized, Double Blind, Placebo-Controlled Phase II Study to Evaluate the Safety, Tolerability, and Activity of Intravenous MLDL1278A in Patients on Standard-of-Care Therapy for Stable Atherosclerotic Cardiovascular Disease (GLACIER - Goal of Oxidized Ldl and Activated Macrophage Inhibition by Exposure to a Recombinant Antibody)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Activity of Intravenous MLDL1278A in Patients on Standard-of-Care Therapy for Stable Atherosclerotic Cardiovascular Disease (GLACIER)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LDL4758g; GC01314 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis
Keywords: BI-204
MeSH Terms: conditions — Atherosclerosis | interventions — MLDL1278A; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Experimental)
  Interventions: Drug: MLDL1278A; Drug: statin, stable dose
- B (Experimental)
  Interventions: Drug: MLDL1278A; Drug: statin, stable dose
- C (Placebo Comparator)
  Interventions: Drug: placebo; Drug: statin, stable dose

INTERVENTIONS:
Drug: MLDL1278A — Single intravenous dose
  Arms: A
Drug: MLDL1278A — Repeating intravenous dose
  Arms: B
Drug: placebo — Repeating intravenous dose
  Arms: C
Drug: statin, stable dose — Repeating oral dose

SUMMARY:
This is a Phase II (proof-of-activity), double-blind, placebo-controlled, randomized, multicenter study of MLDL1278A (also known as BI-204) involving patients on standard-of-care therapy for atherosclerotic cardiovascular disease with evidence of vascular inflammation, as quantified by FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of qualifying vessel (carotid or aortic) plaque inflammation
* Documented atherosclerotic vascular disease clinically stable for at least 3 months prior to screening or type 2 diabetes mellitus with elevated cardiovascular risk
* Use of a stable dose of statin therapy for at least 6 weeks prior to screening. Patients must be capable of maintaining statin therapy at a current dose level from screening until the last follow-up visit.
* For patients taking angiotensin-converting enzyme (ACE) inhibitors (ACE-I) or angiotensin-receptor blockers (ARBs), non-statin lipid-modifying therapy, thiazolidinediones, inhaled steroids, or leukotriene modifying agents, use of a stable dose for at least 6 weeks prior to screening and capable of continuing with that dose for the duration of the study

Exclusion Criteria:

* Occurrence of a cardiovascular event < 6 months prior to screening
* Pregnant, planning to become pregnant during the study, or breastfeeding
* Clinically significant abnormal laboratory values or abnormal ECG or vital signs
* History of anaphylactic reactions
* Newly discovered Type 2 diabetes mellitus (T2DM) (prior to study entry) or medical treatment for T2DM started < 3 months prior to study entry
* Use of insulin, corticosteroids (oral, rectal, or injectable), or other immunosuppressive medications
* Current or recent (within 4 weeks prior to screening) infection, including signs, symptoms or serology of any infection, including HIV, hepatitis B or C
* Impaired renal function
* History of malignancy within 2 years prior to screening
* Current life-threatening condition other than vascular disease that may prevent a patient from completing the study
* Use of an investigational drug or biologic within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study medication
* Exposure to substantial radiation within 12 months prior to screening

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in TBR as measured by FDG-PET/CT | Baseline to Week 12

SECONDARY OUTCOMES:
Incidence and severity of adverse events and clinical laboratory abnormalities as a measure of safety and tolerability of MLDL1278A | Throughout study or until early discontinuation
Effects of MLDL1278A on inflammatory and metabolic biomarkers | Throughout study or until early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lehrer-Graiwer, M.D., Study Director — Genentech, Inc.
Locations (20):
- United States (18):
  - Torrance, California
  - Colorado Springs, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Haverhill, Massachusetts
  - Royal Oak, Michigan
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Newington, New Hampshire
  - New York, New York
  - North Massapequa, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Houston, Texas
- Canada (2):
  - Ottawa, Ontario
  - Montreal, Quebec